CLINICAL TRIAL: NCT07015944
Title: Clinical and Cost-effectiveness of an Integrated Psychosocial Care Plan for Comorbid Depression in Breast Cancer Survivors In Pakistan: A Sequential Multiple Assignment Randomised Trial
Brief Title: Moving on After Breast Cancer Trial for Depressed Breast Cancer Survivors in Pakistan
Acronym: Moving On ABC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Sheffield (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Moving On ABC Plus; NIHR205561 (Other Grant/Funding Number: National Institute of Health and care Research (NIHR))
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder (MDD); Breast Cancer Survivor
Keywords: Breast Cancer; LMICs; Depression; Multimorbidity; SMART; Adaptive interventions; Cognitive Behaviour Therapy; Low intensity intervention
MeSH Terms: conditions — Depressive Disorder, Major; Breast Neoplasms; Depression | interventions — abacavir; Antidepressive Agents

STUDY DESIGN:
Intervention Model Description: Sequential, Multiple Assignment, Randomized Trial (SMART). The SMART design allows investigators to evaluate the effects of different intervention options and develop an adaptive approach to better meet participants' needs
Who Masked: Outcomes Assessor
Masking Description: Trial investigators and trial statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive interventions (Experimental): The adaptive interventions include:
  1. Non-specialist delivered Low intensity guided self-help (Khushi and Khatoon)
  2. Moving on After Breast cancer Plus (Moving on ABC Plus)
  3. Standard pharmacological intervention
  Interventions: Other: Non-specialist delivered Low intensity guided self-help (Khushi and Khatoon); Other: Moving on After Breast Cancer (ABC) plus; Drug: Standardised pharmacological treatment (antidepressants); Other: Enhanced Treatment As Usual (E-TAU)
- Enhanced Treatment As Usual (E-TAU) (Other): Participants in this arm will continue to follow their routine visits to healthcare facilities. They will be regularly monitored by trained research team and will be assessed at weeks 6,18,30, and 48. In addition to psychological assessment at each follow-up, this will include information leaflets based on a brief psychoeducational module to educate participants about the risks, symptoms, management, and referral support information for anxiety and depression.
  Interventions: Other: Enhanced Treatment As Usual (E-TAU)

INTERVENTIONS:
Other: Non-specialist delivered Low intensity guided self-help (Khushi and Khatoon) — This is a manualised intervention comprising of 8 chapters. This is being further co-adapted to contexualise this for breast cancer survivours. The original manual is focused on stories of two breast cancer survivors , Mrs Khushi, means happiness) and Khatoon, means woman in Urdu, with depression and anxiety, describing how they help themselves using CBT strategies.
  Arms: Adaptive interventions
Other: Moving on After Breast Cancer (ABC) plus — This is a high intensity manualised intervention consisting of 12 sessions (60-90 minutes). This manual offers practical support and advice on life after breast cancer, managing difficulties, mindfulness, addressing fatigue, understanding the participant's model of illness, improving personal effectiveness and social relationships. The sessions also include therapist delivered psychoeducation using a CBT model of case formulation and goal setting: identification and formulation of predisposing, precipitating, perpetuating and protective factors of depression and/or anxiety, helping participants to identify core beliefs, where necessary, using downward arrow technique, identifying, and challenging unhealthy thinking patterns at the level of core beliefs using cognitive restructuring, and problem-solving techniques
  Arms: Adaptive interventions
Drug: Standardised pharmacological treatment (antidepressants) — Patients will begin 12 weeks of sertraline treatment initiated at a daily dose of 50 mg for the first 4 weeks. After that, flexible titation of sertraline will be permitted, by 50mg increment every 1 to 2 weeks, as clinically indicated and tolerated to a maximum daily dose of 200 mg
  Arms: Adaptive interventions
Other: Enhanced Treatment As Usual (E-TAU) — Participants in this arm will continue to follow their routine visits to healthcare facilities. They will be regularly monitored by trained research team and will be assessed at weeks 6,18,30, and 48. In addition to psychological assessment at each follow-up, this will include information leaflets based on a brief psychoeducational module to educate participants and families about the risks, symptoms, management, and referral support information for anxiety and depression

SUMMARY:
Breast cancer is the most common cancer among women worldwide, and many survivors experience comorbid mental health conditions such as depression and anxiety, which can significantly worsen health outcomes and increase mortality. This large-scale trial in Pakistan aims to evaluate the clinical and cost-effectiveness of a three-stage adaptive intervention to manage depression among breast cancer survivors. Using a Sequential, Multiple Assignment, Randomised Trial (SMART) design, the study will recruit 26,372 participants aged 18 and above who have completed initial breast cancer treatment (surgery and/or chemotherapy or radiotherapy). Participants will be identified through primary care units, outpatient departments, oncology clinics in public hospitals, and charitable organisations across Pakistan. Depression will be screened using the Patient Health Questionnaire PHQ-9, with diagnosis confirmed by the Structured Clinical Interview Schedule of DSM (SCID). Those randomised to the intervention arm will receive adaptive interventions: starting with low-intensity guided self-help, followed by a high-intensity cognitive behavioural therapy-based programme called "Moving On After Breast Cancer Plus" (Moving on ABC Plus), and for non-responders, an additional pharmacological component will be introduced. Participants in both adaptive intervention and enhance usual care groups will be assessed at multiple time points-baseline, 6, 18, 30, and 48 weeks post-randomisation-using validated tools to measure depression (primary outcome), and anxiety, self-esteem, intrusive thoughts, health-related quality of life, satisfaction with services, and health resource use (secondary outcomes). The study will also include qualitative interviews and focus groups discussions with patients, caregivers, healthcare providers, and policymakers to identify barriers and facilitators to implementation and ensure the intervention is both contextually appropriate and scalable.

DETAILED DESCRIPTION:
Problem statement: Breast cancer is the most prevalent cancer among women globally. The comorbidity of mental health conditions, such as depression and anxiety, significantly increases mortality rates in this population. Despite the complex rehabilitation needs of breast cancer survivors, there is limited knowledge on how to provide individualised support effectively.

Aims/Objectives: The overarching aim of this trial is to evaluate the clinical and cost-effectiveness of a three-stage adaptive intervention for co-morbid depression among breast cancer survivors in Pakistan.

Methods: This study will use a Sequential, Multiple Assignment, Randomised Trial (SMART) design to recruit 26,372 breast cancer survivors who have completed initial treatment (surgery and/or radiotherapy or chemotherapy). Participants, aged 18 years and older, will be recruited from primary care units, medical outpatient units, oncology clinics in public hospitals, and charitable organisations across Pakistan. Eligible participants will be screened for Major Depressive Episode (MDE) using the Patient Health Questionnaire (PHQ-9), with a score of 10 or above indicating potential depression. Diagnosis will be confirmed through the Structured Clinical Interview Schedule (SCID). Participants randomised to the intervention arm will receive a three-stage adaptive intervention, progressing through the following levels based on response: First adaptive intervention - Low-intensity guided self-help. Second adaptive intervention - High intensity "Moving On After Breast Cancer Plus" (Moving on ABC Plus), incorporating Cognitive Behavioural Therapy (CBT). Third adaptive intervention - Moving on ABC Plus combined with pharmacological intervention. All participants, regardless of randomisation, will be assessed at baseline, 6-, 18-, 30-, and 48-weeks post-randomisation using standardised questionnaires to measure: Primary outcome: Depression. Secondary outcomes: Anxiety, self-esteem, intrusive thoughts, health-related quality of life, satisfaction with services, and resource utilisation. Additionally, in-depth interviews and focus group discussions (FGDs) will be conducted with multiple stakeholders-including healthcare providers, policymakers, patients, and caregivers-to explore barriers and facilitators of intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 18 years and above
* Diagnosed with breast cancer (any stage)
* Completed initial treatment (i.e., surgery and/or radiotherapy or chemotherapy) for breast cancer (even if they are currently on hormonal therapy post-initial treatment)
* Total score of 10 or above on the Patient Health Questionnaire (PHQ-9)
* Diagnosis of current Major Depressive Episode (MDE) confirmed using the Structured Clinical Interview for DSM-5 (SCID).

Exclusion Criteria:

* Lacking capacity to provide informed consent, such as those identified by clinicians as having intellectual disabilities, dementia, or severe medical and/or psychiatric illnesses requiring hospitalisation
* Unable to engage in assessments or interventions, including those with stage 4 breast cancer experiencing significant symptoms (e.g., metastatic lesions in the lungs, liver, or bones requiring daily treatment for symptomatic relief, such as the daily use of two or more painkillers), which restrict their capacity to participate
* Currently receiving psychological therapy or taking antidepressant medications (e.g., SSRIs, SNRIs, or other prescribed antidepressants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 26376 (Estimated)
Dates: Start 2025-06-13 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Change in total score from baseline to week 48
  Primary outcome will be depression remission at 48 weeks. This is a 17 item, clinician administered assessment measure to assess severity of depressive symptoms over past week. Total score of 0-7 is considered as "normal" (clinical remission), and a total score of 20 or higher is considered as moderate to severe.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder | Change in Total Score from baseline to week 6, 18, 30 and 48
  Severity of anxiety over last two weeks will be assessed using the Generalized Anxiety Disorder - 7 . Individuals with total score between 0 to 4 will be categories as having "minimal anxiety", 5 to 9 "mild anxiety", 10 to 14 "moderate anxiety" and 15 to 21 "severe anxiety".
EuroQol-5 Dimensions | Change in total score from baseline to week 6, 18, 30 ans 48
  Health-related quality of life will be assessed using the EQ-5D. This questionnaire assesses quality of life by exploring 5 areas: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is rated as one of the followings: no problems, slight problems, moderate problems, severe problems and extreme problems. Higher score indicate better quality of life. The range for EQ-5D scores is between -0.594 and 1, where 1 signifies full health. Scores below 0 indicate health states worse than death.
Functional Assessment of Cancer Therapy - Breast | Change in total score from baseline to week 6, 18, 30 and 48
  This scale measures health-related quality of life in breast cancer patients in five domains: physical, social, emotional, functional well-being as well as a breast-cancer sub-scale Higher score indicate better quality of life. Minimum possible score on this scale is 0 and maximum possible score is 144.
Rosenberg Self Esteem Scale | Change in total score from baseline to week 6, 18, 30 and 48
  Self-esteem will be assessed using this scale. Total score on the scale ranges from 0-30. Total score between 15 to 25 is considered as within normal range and total score below 15 is indicative of low self-esteem
Multidimensional Scale for Perceived Social Support | Change in total score from baseline to week 6, 18, 30 and 48
  This scale aims to assess an individual's perception of support from 3 sources: family, friends and a significant other. Total score between 12 to 35 is categorised as "low perceived support", 36 to 60 "medium perceived support", and 61 to 84 "high perceived support".
Client Satisfaction Questionnaire | Change in total score from baseline to week 6, 18, 30 and 48.
  Satisfaction with treatment/services will be assessed using this scale. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Client Service Receipt Inventory | Change in score from baseline to week 6, 18, 30 and 48
  Information on participants' use of both formal and informal (such as Imams/faith healers) health services was collected at baseline and follow-up assessments using a structured form.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, MD, Principal Investigator — Pakistan Institute of Living and Learning
Locations (1):
- Pakistan Institute of Living and Learning, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized data will be shared. Requests to be made to Principal Investigator
Supporting Information: Study Protocol
Time Frame: Once the trial results are published
Access Criteria: Requests should be made to Principal Investigator